CLINICAL TRIAL: NCT01318486
Title: HepZero:Heparin Free Dialysis With Evodial: A Prospective Multicenter, Open, Randomized, Controlled Clinical Study With Parallel Groups
Brief Title: HepZero:Heparin Free Dialysis With Evodial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Statistical Analysis : CIC CHU Brabois Nancy (Unknown); Gambro Lundia AB (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1483
Record Dates: First submitted 2011-03-11; First posted 2011-03-18 (Estimated); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Disease; Patients Requiring Heparin Free Dialysis Treatments
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heparin free dialysis standard of care (Active Comparator): Standard of care: can be either saline flushes or predilution (on-line or bags)
  Interventions: Other: Heparin free dialysis technique
- Heparin free dialysis with Evodial (Experimental)
  Interventions: Device: Evodial

INTERVENTIONS:
Other: Heparin free dialysis technique — Saline flushes or predilution
  Other Names: Standard of care
  Arms: Heparin free dialysis standard of care
Device: Evodial — Evodial dialyer
  Arms: Heparin free dialysis with Evodial

SUMMARY:
The study hypothesis is that with Evodial in patients requiring heparin free dialysis, the heparin free treatment can be performed easily (without saline flushes or blood predilution) and is at least not inferior and maybe superior to the standard care heparin free treatment in terms of clotting.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring heparin free dialysis treatments on nephrologists' prescription,
* Chronic ESRD patients treated by maintenance hemodialysis for at least 3 months,
* Patients with a well functioning blood access that can allow a blood flow of at least 250 ml/min,
* Patients aged 18 years or more,
* Written consent to participate in the study (informed consent).

Exclusion Criteria:

* Patients in ICU settings,
* AKI patients,
* Patients dialyzed in self care, satellite HD units,
* Patients treated in single needle mode,
* Known heparin contraindication (HIT type II),
* Patients requiring blood and other labile blood products (i.e. fresh frozen plasma, platelets, etc …) transfusion during hemodialysis treatment,
* Patients receiving oral anticoagulants (including Anti vitamin K),
* Patients receiving a combination of anti-platelets agents,
* Patients treated with unfractionated or low molecular weight heparin beside the dialysis treatment to prevent deep vein thrombosis,
* Pregnant/ planning pregnancy and lactating women during study period,
* Adult patients protected by the law,
* Patients are not affiliated to health insurance system (beneficiary or dependant)
* Participation in other interventional studies during the study period,
* Patients that have already been included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 265 (Actual)
Dates: Start 2011-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Clotting of the dialysis session | During first dialysis session_Dialysis duration: 4 hours
  To evaluate the rate of successful treatments, clotting in the air traps will be evaluated using a scale grading from 1 to 4 and previously described in the literature.
  The first heparin free dialysis treatment will be considered successful when there is:
  * No complete occlusion of air traps or dialyzer rendering dialysis impossible (grade 4 of the scale),
  * No additional saline flushes to prevent clotting,
  * No change of dialyzer or blood lines because of clotting
  * No premature stop (early rinse-back) because of clotting

SECONDARY OUTCOMES:
Clotting during consecutive dialysis session | 2nd and 3rd consecutive dialysis sessions
  As for the first heparin free dialysis treatment, treatments will be considered successful when there is :
  * No complete occlusion of air traps or dialyzer rendering dialysis impossible (grade 4 of the scale),
  * No additional saline flushes to prevent clotting,
  * No change of dialyzer or blood lines because of clotting
  * No premature stop (early rinse-back) because of clotting.
Follow up of clotting during the dialysis sessions | During all dialysis sessions
  * Grade 1: No detectable clotting
  * Grade 2: Minimal clot formation (Presence of fibrinous ring)
  * Grade 3: Clot formation (up to 5 cm) but dialysis still possible
  * Grade 4: complete occlusion of air traps or dialyzer rendering dialysis impossible
Efficacy: Ultrafiltration | During all dialysis sessions
  Measurement of urea, creatinine and ionogramm, UF achieved
Ease of use | During all dialysis sessions
  Collection of saline flushes performed (volume and time)
Incidence of AEs/SAEs | During all dialysis sessions
  Follow-up of AEs/SAEs

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Laville, Pr, Study Chair — CHU Edouard Herriot Lyon
Locations (10):
- Erasme Hospital, Brussels, Belgium
- George Dumont Hospital, Moncton, New Brunswick, Canada
- France (3):
  - CHU Edouard Herriot, Lyon
  - CHU Brabois, Nancy
  - CHU de Saint-Étienne - Hôpital Nord, Saint-Priest-en-Jarez
- UMCG, Groningen, Netherlands
- Gdanski Uniwersytet Medyczny, Gdansk, Poland
- Spain (2):
  - Hospital Universitary German Trias i Pujol, Badalona
  - Vall d'Hebron Hospital, Barcelona
- Royal Liverpool University Hospital, Liverpool, United Kingdom

REFERENCES:
- [Background] Kim YG. Anticoagulation during haemodialysis in patients at high-risk of bleeding. Nephrology (Carlton). 2003 Oct;8 Suppl:S23-7. doi: 10.1046/j.1440-1797.8.s.3.x. PMID 15012687
- [Background] European Best Practice Guidelines Expert Group on Hemodialysis, European Renal Association. Section V. Chronic intermittent haemodialysis and prevention of clotting in the extracorporal system. Nephrol Dial Transplant. 2002;17 Suppl 7:63-71. doi: 10.1093/ndt/17.suppl_7.63. No abstract available. PMID 12386229
- [Background] Chanard J, Lavaud S, Maheut H, Kazes I, Vitry F, Rieu P. The clinical evaluation of low-dose heparin in haemodialysis: a prospective study using the heparin-coated AN69 ST membrane. Nephrol Dial Transplant. 2008 Jun;23(6):2003-9. doi: 10.1093/ndt/gfm888. Epub 2007 Dec 21. PMID 18156457
- [Background] Lohr JW, Schwab SJ. Minimizing hemorrhagic complications in dialysis patients. J Am Soc Nephrol. 1991 Nov;2(5):961-75. doi: 10.1681/ASN.V25961. PMID 1760540
- [Background] Yixiong Z, Jianping N, Yanchao L, Siyuan D. Low dose of argatroban saline flushes anticoagulation in hemodialysis patients with high risk of bleeding. Clin Appl Thromb Hemost. 2010 Aug;16(4):440-5. doi: 10.1177/1076029609334628. Epub 2009 Oct 14. PMID 19833621
- [Derived] Natale P, Palmer SC, Ruospo M, Longmuir H, Dodds B, Prasad R, Batt TJ, Jose MD, Strippoli GF. Anticoagulation for people receiving long-term haemodialysis. Cochrane Database Syst Rev. 2024 Jan 8;1(1):CD011858. doi: 10.1002/14651858.CD011858.pub2. PMID 38189593
- [Derived] Laville M, Dorval M, Fort Ros J, Fay R, Cridlig J, Nortier JL, Juillard L, Debska-Slizien A, Fernandez Lorente L, Thibaudin D, Franssen C, Schulz M, Moureau F, Loughraieb N, Rossignol P. Results of the HepZero study comparing heparin-grafted membrane and standard care show that heparin-grafted dialyzer is safe and easy to use for heparin-free dialysis. Kidney Int. 2014 Dec;86(6):1260-7. doi: 10.1038/ki.2014.225. Epub 2014 Jul 9. PMID 25007166
- [Derived] Rossignol P, Dorval M, Fay R, Ros JF, Loughraieb N, Moureau F, Laville M. Rationale and design of the HepZero study: a prospective, multicenter, international, open, randomized, controlled clinical study with parallel groups comparing heparin-free dialysis with heparin-coated dialysis membrane (Evodial) versus standard care: study protocol for a randomized controlled trial. Trials. 2013 Jun 1;14:163. doi: 10.1186/1745-6215-14-163. PMID 23725299